CLINICAL TRIAL: NCT00847314
Title: Efficacy and Tolerability of Testogel® / Nebido in Combination With a Standardised Exercise and Diet Programme in Hypogonadal Male Patients With Abdominal Obesity Compared With Exercise and Diet Programme
Brief Title: Efficacy and Tolerability of Testogel/Nebido in Combination With Exercise and Diet in Hypogonadal Male Patients
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Schering Pharma AG
Other Study IDs: 13899; NE0602 (Other: Other company ID)
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Abdominal obesity; Physical exercise; Testosterone
MeSH Terms: conditions — Hypogonadism; Obesity, Abdominal; Motor Activity | interventions — Testosterone Propionate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Testosterone Undeconate (Nebido-R, BAY86-5037)

INTERVENTIONS:
Drug: Testosterone Undeconate (Nebido-R, BAY86-5037) — Male patients > 35yrs in medical practices fulfilling all criteria for documentation.

SUMMARY:
With advancing age testosterone levels decline in men. Low testosterone levels plus certain symptoms are called "Late Onset Hypogonadism (LOH)". Adipose tissue may contribute to testosterone deficiency. On the other hand testosterone deficiency again leads to a decrease in lean body mass and an increase in fat mass - one of the clinical signs / symptoms of LOH. Lifestyle changes (diet, exercise) alone or in combination with testosterone replacement (TRT), have an influence on the symptoms of LOH. The aim of this study is to assess the additional impact of TRT on Aging Male Symptom Score (AMS) and adiposity (waist circumference) in patients, who are on a diet and exercise program.

ELIGIBILITY:
Inclusion Criteria:

* Male patients > 35yrs
* Waist Circumference > 102cm
* Clinically and biochemically confirmed hypogonadism (testosterone group)
* Willingness to attempt weight optimization

Exclusion Criteria:

* Androgen dependent carcinoma of the prostate or male mammary gland, past or present history of liver tumours
* hypersensitivity towards the active pharmaceutical ingredient or other ingredients.

Ages: 35 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male patients in medical practices > 35yrs fulfilling all criteria for documentation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Waist Circumference | At each visit

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany